CLINICAL TRIAL: NCT02727842
Title: Usability of the CP950 Sound Processor With Experienced Cochlear Implant Users
Brief Title: Usability of the CP950 Sound Processor
Acronym: C950
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5657
Record Dates: First submitted 2016-03-17; First posted 2016-04-05 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Hearing Loss
Keywords: cochlear implant; Sound Processor
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment group (Experimental): All patients will receive the CP950 Sound Processor and be part of the treatment group for one month which is programmed via the wireless programming pod
  Interventions: Device: CP950 Sound Processor; Device: Wireless programming pod

INTERVENTIONS:
Device: CP950 Sound Processor — An off-the-ear processor configuration with identical functionality to the commercially approved CP910/920 processor
Device: Wireless programming pod — The CP950 Sound Processor will be programmed by the wireless programming pod, which is needed as the interface to commercially approved programming software

SUMMARY:
Studying usability and gaining feedback of the CP950 Sound Processor in experienced cochlear implant recipients.

DETAILED DESCRIPTION:
One month protocol, with 2 study visits. The aim of the study to is to gain patient and audiologist feedback on their experience and usability with the device and wireless programming pod.

ELIGIBILITY:
Inclusion Criteria:

1. At least 6 months experience with a Nucleus 24 series or later implant in at least one implanted ear
2. Subjects age 12 and older who are cognitively and developmentally able to complete all study related questionnaires as deemed by the principal investigator or delegated staff
3. At least 3 months experience with the CP810,CP920 or CP910 sound processor
4. Ability to use 2 zinc air batteries with their current program (MAP)
5. Willingness to participate in and to comply with all requirements of the protocol for the duration of the trial

Exclusion criteria:

1. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and prosthetic device
2. Additional disabilities that would prevent participation in evaluations
3. Implant types not currently supported by the CP950 sound processor (i.e.,N22)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rocky Mountain Ear Center, Englewood, Colorado
  - NYU, New York, New York
  - Hearts for Hearing, Oklahoma City, Oklahoma

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Sound processor per participant
Period: Overall Study
Arm/Group | Treatment Group
Started | 30; 1 Sound processor per participant
Completed | 30; 1 Sound processor per participant
Not Completed | 0; 0 Sound processor per participant

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 18
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction Through Usability of the CP950 Sound Processor as Measured by the CP950 Take Home Questionnaire
Description: To evaluate usability of the CP950 sound processor using the CP950 Take Home Questionnaire for existing cochlear implant users.
  Specifically:
  1. Patient Reported Hearing Performance
  2. Retention & Comfort
  3. Ease of use
  4. Use of remote controls
  5. Look & feel
  6. Reliability
  7. Maintenance & use
Time Frame: 1 month
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: All study participants were analyzed in the treatment group.
Arm/Group | All Subjects
Number analyzed (Participants) | 30
Participants
  Satisfiaction with retention accessory | 22
  Satisfaction with hearing performance | 28
  Agreed sound processor is comfortable | 27
  Agreed sound processor is easy to use | 28
  Satisfied with look and feel of processor | 27
  Agreed sound processor was reliable | 29
  Agreed sound processor is easy to clean | 24

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were no unanticipated or serious adverse events reported. The All-Cause Mortality rate was zero.
Groups:
- Treatment Group: There were no unanticipated or serious adverse events reported. The All-Cause Mortality rate was zero.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=30)
Mircrophone housing (Product Issues) | 1 (1) — Intermittent sound processor. The adverse event was resolved by replacing the processor. The device was subsequently analyzed and found to have dislodged microphones from the housing.
Skin flap (Product Issues) | 1 (1) — Infection or swelling at implant site. August 30, 2016 was reported date of onset, and reported to the clinic on September 3, 2016. The adverse event was resolved on September 6, 2016 by antibiotic treatment.

LIMITATIONS AND CAVEATS:
Short-term usability study, in a small population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT02727842/Prot_001.pdf